CLINICAL TRIAL: NCT05010187
Title: Preventing Alcohol Misuse and Consequences in Vulnerable Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23AA028513 (NIH); K23AA028513 (NIH)
Record Dates: First submitted 2021-07-20; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Motivational Interview (MI) (Experimental): Participants will complete a brief motivational interview focusing on determinants of women's alcohol use, including a focus on normative perceptions as well as motives for drinking.
  Interventions: Behavioral: Behavioral: Motivational Interview (MI)
- Behavioral: Health Coaching (HC) (Active Comparator): Participants will complete a brief health coaching interview and session focusing on educational modules.
  Interventions: Behavioral: Behavioral: Health Coaching (HC)

INTERVENTIONS:
Behavioral: Behavioral: Motivational Interview (MI) — Single-session, brief motivational interview.
  Arms: Behavioral: Motivational Interview (MI)
Behavioral: Behavioral: Health Coaching (HC) — Single-session health coaching.
  Arms: Behavioral: Health Coaching (HC)

SUMMARY:
Heavy alcohol use is a pressing public health issue that results in more negative consequences for young adult women, despite them drinking at lower rates than their male peers. However, particular groups of women, such as women who identify as lesbian and bisexual (i.e., sexual minority women), evidence markedly higher rates of alcohol misuse as well as negative consequences from this use. Sexual minority women are more likely to use alcohol, do so at problematic levels, and to meet criteria for alcohol use disorders than heterosexual women and sexual minority men. Despite these disparities, as well as evidence that sexual minority women have unique mechanisms of risk (e.g., minority stress, social context), there are currently no interventions designed to reduce alcohol misuse among sexual minority women. This study represents the first attempt to design an in-person intervention specifically tailored to sexual minority women, which will be accomplished through an Intervention Mapping framework to identify behavioral determinants of their use (e.g., minority stress and distress; social context) and then map effective behavior change strategies onto these determinants.

DETAILED DESCRIPTION:
This particular study aim is devoted to the piloting of a brief motivational intervention to reduce alcohol misuse and consequences among sexual minority women. The objective of this study aim is to examine the preliminary feasibility and acceptability of the intervention following treatment development and refinement. Participants will be randomized to a brief intervention or an attention-matched control arm. Participants in both conditions will complete: a baseline survey as well as a follow-up assessment at 1- and 4-months post-intervention. The investigators hypothesize that the developed intervention will be feasible (as indicated by the number of women eligible who consent, attend their intervention session, and return for follow up). The investigators also hypothesize that the intervention will be acceptable to sexual minority women. The investigators will also obtain preliminary evidence of intervention efficacy in terms of alcohol use outcomes. Specifically, the investigators hypothesize that participants in the intervention will report less frequent heavy episodic drinking and fewer alcohol consequences post-intervention compared with those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* English speaking;
* Currently reporting heavy drinking;
* Identifies as a sexual minority woman.

Exclusion Criteria:

* Unwilling or unable to provide informed consent;
* Low literacy (i.e., reporting they "often" or "always" need someone to read instructions, pamphlets, or other written material from a doctor or pharmacy to them)
* Women who report intention to move away during study period.
* Active suicidality.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Identifies as a woman.
Enrollment: 70 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | Through study completion, an average of 4 months
  Rates of enrolling after eligibility; attendance after randomization
Acceptability of Intervention | Immediately post-intervention
  Self-reported acceptability of the intervention. Adequate acceptability will be defined as ≥ 80% endorsement of being at least somewhat satisfied with participation.

SECONDARY OUTCOMES:
Alcohol use quantity | Through study completion, an average of 4 months
  Typical number of drinks per week.
Alcohol consequences | Through study completion, an average of 4 months
  Self-report measure of level of alcohol-related consequences experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa L Norris, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No